CLINICAL TRIAL: NCT07067658
Title: Monitoring Oedema in Heart Failure to Improve Function and Reduce Hospitalisation Risk
Acronym: ME-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heartfelt Technologies (Industry)
Collaborators: Manchester University NHS Foundation Trust (Other Government); University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HFT-2025-1
Record Dates: First submitted 2025-07-04; First posted 2025-07-16 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
Keywords: Peripheral Oedema; Heart Failure Decomposition; Heart Failure Hospitalization
MeSH Terms: conditions — Heart Failure | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: This 12-month study involves up to 300 patients using the Heartfelt device at home.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both participants and care providers will be blinded, thus will not know whether patients are in the control or intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Standard Care + Heartfelt Device (Experimental): Heartfelt device's camera-based system passively measures foot and leg swelling each day as participants walk past it. Patients in this experimental control arm will not receive health alerts from the Heartfelt device, though data will still be passively collected.
  Patients will also be provided with the British Heart Foundation patient booklet to improve their understanding and self-monitoring of the disease.
  Interventions: Device: Installation of Heartfelt Device; Other: Enhanced Standard care; Other: Questionnaires; Device: Heartfelt device alerting system
- Enhanced Standard Care (Control) (Active Comparator): In addition to standard care activities, participants have the Heartfelt device at home. During this arm, data is captured without sending health alerts or measurement data to the patient, carers and clinicians.
  Patients will also be provided with the British Heart Foundation patient booklet to improve their understanding and self-monitoring of the disease.
  Interventions: Device: Installation of Heartfelt Device; Other: Enhanced Standard care; Other: Questionnaires

INTERVENTIONS:
Device: Installation of Heartfelt Device — Device installed in the patient's home and capturing foot volume data which are processed in the cloud.
  Other Names: Remote Patient Monitoring Device
Other: Enhanced Standard care — Patients with heart failure are advised to weigh daily and to report weight increase to their clinician. They should also report changes in breathlessness, tiredness and other symptoms associated with heart failure decompensation. At the start of the study, they will be reminded (or told) about the importance of self-checks and will be handed a patient booklet (from the British Heart Foundation) to standardise patients' knowledge.
  Other Names: Daily Weighing; Breathlessness; Dizziness; Tiredness
Other: Questionnaires — Patients are presented with one or more optional questionnaires (some validated, some bespoke)
  Other Names: 5Q-5D; Bespoke Questionnaires
Device: Heartfelt device alerting system — The Heartfelt device sends alerts on the active comparator arm to the patients directly (audio-visual alert on the device, and app alerts), carers and/or medical professionals.
  Other Names: Remote patient monitoring device
  Arms: Enhanced Standard Care + Heartfelt Device

SUMMARY:
This study will evaluate the Heartfelt device, a novel, passive monitoring system that detects early signs of fluid build-up in patients (oedema) with heart failure by measuring changes in foot and lower leg volume through capture of 3D images. The trial will assess whether this device, when added to standard NHS care, improves quality of life and reduces heart failure-related events compared to standard care alone.

DETAILED DESCRIPTION:
Heart failure often causes fluid build-up in the legs and lungs, leading to symptoms like swelling and breathlessness. Spotting these signs early is important to help prevent worsening health and hospital admissions. While patients are encouraged to monitor their weight and symptoms, this can be hard to keep up with.

The study will involve 300 participants from at least 15 NHS hospitals and GP practices across the UK. People will be randomly placed into one of two groups: one will receive standard NHS care (including regular weight checks and symptom monitoring), and the other will receive the same care plus the Heartfelt device. The trial is partly blinded: participants may see technical messages (e.g. if the device goes offline), but only the group using the device will trigger clinical alerts.

The Heartfelt device takes daily images of the feet to track changes in size, without the need for any extra effort from the user. If important changes are spotted, alerts are sent to the clinical team so they can act quickly.

The study will look at quality of life, how often the device sends useful data, healthcare use, and how teams respond to alerts. It will also explore how easy the device is to use and whether it offers good value for money.

Patients will help shape the study to make sure the findings are relevant and useful for future care.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years
* Diagnosis of heart failure (any aetiology or left ventricular ejection fraction classification), any timeframe
* Currently prescribed ≥40 mg/day of furosemide (or equivalent loop diuretic) for at least one month.
* Heart failure hospital admission and moderate or severe leg oedema in the previous 12 months.
* Lives in the UK, with a home environment suitable for installation of the Heartfelt device.

Exclusion Criteria:

* Amputation of both feet
* Bed-bound for more than 20h per 24h period
* Bandages to lower limbs every day
* Regular wheelchair user inside their home
* No fixed abode
* Participation in another interventional trial that may interfere with endpoints
* Life expectancy <6 months, in the opinion of the investigator
* Inability to provide informed consent due to cognitive impairment
* Language barriers that preclude understanding of trial procedures (unless translation resources are available in relevant language)
* Inability to install the device (even with assistance) allowing at least 6 months of data capture by the end of the study.
* Patients with severe aortic stenosis or awaiting a heart procedure or surgery
* Patient with end stage renal disease (eGFR <20)
* Pregnancy or lack of contraceptive measures if of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Composite Clinical Events | Over 12-months period.
  Unplanned hospital attendance (clinic, emergency, or admission) or death due to heart failure, cardiovascular, respiratory, or renal causes. Recurrent events will be included and adjudicated, providing a comprehensive measure of clinical deterioration over 12 months.
Health-Related Quality of Life (EQ-5D-5L) | Collected at baseline, 3, 6, 9, and 12 months
  Patient-reported quality of life measured using EQ-5D-5L, collected at baseline and follow-up (3, 6, 9, 12 months), with primary analysis at 12 months. This validated instrument captures overall health status across five domains and includes a visual analogue scale.
  * Measured using the EQ-5D-5L index
  * Collected at baseline, 3, 6, 9, and 12 months.
  * Primary time point: 12 months.
  EQ-5D-5L responses will be converted to utility scores on a scale from -0.59 to 1, where 1 represents the best health state, using the UK EQ-5D-5L value set. Patients with at least two or more utility scores during follow-up will be included in the analysis.

SECONDARY OUTCOMES:
Days Lost to Hospitalisation or Death | Over 12-months period.
  Total number of days lost due to hospitalisation for cardiovascular, respiratory, or renal conditions, or due to all-cause mortality.
Daily Data Availability | Over 12-months period.
  Proportion of days with successful data capture from the Heartfelt device and weighing scales, based on device-generated records or contemporaneous self-report.
Guideline-Recommended Medication Score | Over 12-months period.
  Adherence to guideline-recommended heart failure medications will be assessed using a guideline-recommended medication score, calculated at 3, 6, 9, and 12 months and averaged across these time points. The score is based on the number of eligible medication classes prescribed, with 1 point assigned per class (e.g., ACEi/ARB/ARNI, beta-blocker, mineralocorticoid receptor antagonist [MRA]). The score ranges from 0 to 3, with 3 being the optimal medication score.
  The score is adjusted for patient eligibility: will be calculated only for patients with heart failure with reduced ejection fraction (HFrEF).
All-Cause Hospitalisations | Over 12-months period.
  Number of hospitalisations from any cause, analysed as recurrent events and adjusted for the competing risk of death.
Loss of Independence or Mortality | During the 12-month trial period.
  Composite measure of new admission to a long-term care facility or all-cause mortality.
Death and Cause of Death | During 12-months trial period.
  Classification of all deaths recorded during the trial as heart failure-related, other cardiovascular, or non-cardiovascular causes, based on clinical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Croydon Health Services NHS Trust, Croydon, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will only be shared if approved by the Trial Management Group and that suitable ethics approvals has been received for sharing of such information.